CLINICAL TRIAL: NCT02051101
Title: Pathogenic Mechanisms of Port Wine Stain and Repository of Port Wine Stain Biopsy Samples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Wenbin Tan, Ph.D. Project Scientist, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20139396
Record Dates: First submitted 2013-11-06; First posted 2014-01-31 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Port Wine Stain Birthmark (Other): Biopsy sample from Port Wine Stain Birthmark
  Interventions: Other: Biopsy sample from Port Wine Stain Birthmark

INTERVENTIONS:
Other: Biopsy sample from Port Wine Stain Birthmark — Biopsy sample from Port Wine Stain Birthmark

SUMMARY:
The purpose of this study is to investigate the pathogenic mechanisms of Port Wine Stain, collect biopsy samples and blood samples to characterize exosomes and metabolites from Port Wine Stain.

DETAILED DESCRIPTION:
The researcher can detect the defects in nervous system innervation to cutaneous blood vessels contribute to the pathogenesis of Port Wine Stain . Unveiling the pathogenic mechanisms of PWS is crucial to the design of new therapeutic strategies and can use the results to improve current PWS therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of all ages.
* Not pregnant.
* Has diagnosis of port wine stain on the arms, legs, chest, bac.
* Ability to understand and carry out subject instructions.
* Subject willing to have skin biopsies on port wine stain and normal skin areas.

Exclusion Criteria:

* Pregnant women.
* Port Wine Stain on the face.
* History of skin cancer.
* Current participation in an investigational drug evaluation
* Concurrent use of known photosensitizing drugs.

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Characterization of Port Wine Stain Birthmark tissue sample | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John s Nelson, MD, Study Director — Beckman Laser Institute, UCI; Winbin Tan, PhD, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute, Irvine, California, United States